CLINICAL TRIAL: NCT00303420
Title: Alteplase for Blood Flow Restoration in Hemodialysis Catheters: A Randomized Prospective Clinical Trial
Brief Title: Alteplase for Blood Flow Restoration in Hemodialysis Catheters
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to enrol enough people to achieve the full sample size
Sponsor: University of Manitoba (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Lavern M. Vercaigne, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2003:119
Record Dates: First submitted 2006-03-15; First posted 2006-03-16 (Estimated); Last update posted 2008-12-19 (Estimated); Status verified 2008-12

CONDITIONS: Thrombosis
Keywords: catheter; hemodialysis; dysfunction; thrombolytic; alteplase
MeSH Terms: conditions — Thrombosis | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Alteplase used by normal dwell procedure
  Interventions: Drug: alteplase dwell arm
- 2 (Experimental): Alteplase given by an new "push" protocol
  Interventions: Drug: Alteplase "push" protocol

INTERVENTIONS:
Drug: Alteplase "push" protocol — alteplase 2 mg / lumen. Instill and wait 10 minutes, instill 0.3 ml normal saline, wait 10 minutes, instill 0.3 ml of normal saline, wait 10 minutes and aspirate.
  Other Names: CathFlo; alteplase; rTPA
  Arms: 2
Drug: alteplase dwell arm — alteplase 2 mg / lumen. Instill and let it dwell for 30 minutes. Assess catheter and allow to dwell for a total of 2 hours if necessary
  Other Names: Cathflo; alteplase; rTPA
  Arms: 1

SUMMARY:
We are investigating a new way of administering alteplase to remove clots from hemodialysis catheters. Currently, alteplase is left to dwell inside the catheter between dialysis treatments to dissolve the clot and restore blood flow through the catheter. We have developed a new way to administer alteplase by advancing it to the tip of the catheter at regular 10 minute intervals. We hypothesize that our new "push" protocol will dissolve clots in hemodialysis catheters better and faster than the current dwell method.

DETAILED DESCRIPTION:
Central venous catheters are commonly used for vascular access in the hemodialysis population. A common complication is low / no blood flow through the catheter due to clots. These are serious situations because patients may miss dialysis sessions and suffer significant morbidity. In an attempt to dissolve the clots and restore blood flow, thrombolytics are frequently instilled into the catheters between dialysis sessions . However, we have developed and new "push" protocol that advances fresh thrombolytic (alteplase) to the tip of the catheter in order to facilitate more effective and faster removal of the clot. We hypothesize that our new "push" protocol will dissolve clots in hemodialysis catheters better and faster than the current dwell method.

ELIGIBILITY:
Inclusion Criteria:

1. Adults > 18 yrs old
2. Hemodialysis patients
3. Vascular access with a permanent catheter
4. No prior rt-PA use in the catheter over the previous 21 days
5. One rt-PA instillation per catheter (i.e. we will only document the results of 1 rt-PA instillation per catheter. Numerous rt-PA instillations in the same catheter will NOT be considered new events, and not entered into the study)

Exclusion Criteria:

1. Critically ill patients in the ICU setting.
2. Contraindications / cautions with alteplase use including: known hypersensitivity to alteplase or its components (l-arginine, phosphoric acid, polysorbate 80), patients with known conditions associated with bleeding events (e.g.intracranial bleed in last 4 weeks, major hemorrhage in last 4 weeks (Hgb drop of 20 g/L)), recent surgery (<48 hours), recent biopsy (<48 hours), hemostatic defects including severe hepatic disease, or current intracranial / intraspinal neoplasm.
3. Hemodialysis catheter has been in the patient less than 14 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2004-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with pre-thrombolytic blood flows less than 200 ml/min achieving a "sustainable" post thrombolytic blood flow > or = 300 ml/min. | 4 hours

SECONDARY OUTCOMES:
Highest recorded "sustainable" blood flow (ml/min) pre- and post- thrombolytic administration. | 4 hours
Change in Kt/V from the treatment before thrombolytic administration compared to the treatment after thrombolytic administration. | 72 hours
Change in "litres processed / time" from the treatment before thrombolytic administration compared to the treatment after thrombolytic administration. | 72 hours
Serious adverse events including major bleeding within 24 hours of alteplase administration | 30 days post-last dose

CONTACTS AND LOCATIONS:
Overall Officials: Lavern M Vercaigne, Pharm.D., Principal Investigator — University of Manitoba; James M Zacharias, MD, Principal Investigator — University of Manitoba, Internal Medicine, Section of Nephrology
Locations (9):
- Canada (9):
  - Brandon General Hospital, Brandon, Manitoba
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Seven Oaks Hospital, Winnipeg, Manitoba
  - Health Sciences Centre, Winnipeg, Manitoba
  - St. Joseph's Hospital, Hamilton, Ontario
  - Grand River Hospital, Kitchener, Ontario
  - Thunderbay Regional Health Sciences Centre, Thunderbay, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Maisonneuve Rosemont Hospital, Montreal, Quebec

REFERENCES:
- [Background] Zacharias JM, Weatherston CP, Spewak CR, Vercaigne LM. Alteplase versus urokinase for occluded hemodialysis catheters. Ann Pharmacother. 2003 Jan;37(1):27-33. doi: 10.1345/aph.1C105. PMID 12503929